CLINICAL TRIAL: NCT06708650
Title: A Single-arm, Single-center, Open-label Study to Evaluate the Efficacy and Safety of SFRT Combined With PD-1 Inhibitors and Anti-VEGFR in Unresectable Hepatocellular Carcinoma
Brief Title: Combination of SFRT, PD-L1 Inhibitor, and Anti-VEGF in Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guiping People's Hospital (Other)
Responsible Party: Principal Investigator, Yaocan Xu, associate chief physician, Youjiang Medical College for Nationalities
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GuipingPH-HCC-SFRT
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma; Radiotherapy; PD-1 Inhibitors
Keywords: Hepatocellular Carcinoma; radiotherapy; PD-1 Inhibitors; SFRT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of SFRT, PD-L1 inhibitor, and Anti-VEGF in Advanced Hepatocellular Carcinoma (Experimental): Combination of SFRT, PD-L1 inhibitor, and Anti-VEGF in Advanced Hepatocellular Carcinoma
  Interventions: Radiation: Combination of SFRT, PD-L1 inhibitor, and Anti-VEGF

INTERVENTIONS:
Radiation: Combination of SFRT, PD-L1 inhibitor, and Anti-VEGF — Patients received intravenous PD-1 inhibitor 200mg(Camrelizumab, Tislelizumab, or Sintilimab) plus oral Apatinib 250 mg or Lenvatinib 12mg (for bodyweight ≥60 kg) or 8 mg/kg (for bodyweight <60 kg) daily, and additional SFRT for primary liver tumor. PD-1 inhibitor is administered for 2 years or until disease progression or intolerance. Anti-VEGFR is continued until disease progression or intolerance. SFRT implementation plan is as follows: The GTV consists of 2-5 sub-target volumes, which are cylindrical shapes with a diameter of 1.6cm, a height of 2cm, and an interval of 3-5cm. The total volume of the GTV is about 8-20cc, and the distance between the GTV and the OARs is greater than 2cm. The prescribed dosage for each course of radiotherapy is 24 Gy in 3 daily fractions (8Gy x 3F), with a 3-week interval between courses (Q3W). The total courses of radiotherapy shall not be less than 2 (depending on the efficacy and cumulative dose of OARs).

SUMMARY:
PD-1 inhibitor plus anti-VEGFR has become the established standard first-line systemic treatment for unresectable hepatocellular carcinoma (HCC). Despite an improved objective response rate (ORR) of around 30%, the majority of patients face HCC progression and liver failure. Developing a new combined treatment strategy to overcome resistance to anti-PD-L1 and anti-VEGF is essential to improve patient outcomes. Stereotactic radiotherapy (SBRT) can enhance immune response through various mechanisms, and its immunomodulatory effect has been confirmed in multiple solid tumors. However, due to the limitation of the OAR tolerance dose, large-volume tumors are unsuitable for SBRT treatment. To overcome this issue, researchers have introduced the spatially fractionated radiation therapy (SFRT) mode, which allows for a highly uneven radiation dose distribution within the tumor volume. SFRT is an emerging radiotherapy technique with high clinical response rates and low radiation-related toxicity in large-volume solid tumors. Therefore, the investigators conducted this single-arm, single-arm, open-label study to evaluate the efficacy and safety of SFRT combined with PD-1 inhibitors and anti-VEGFR in unresectable HCC. The primary endpoint is objective response rate (ORR), and secondary endpoints include overall survival (OS), progression-free survival (PFS), and toxicity.

DETAILED DESCRIPTION:
This is a single-arm, single-center, open-label study to evaluate the efficacy and safety of SFRT combined with PD-1 inhibitors (Camrelizumab, Tislelizumab or Sintilimab) and anti-VEGFR (Apatinib or Lenvatinib) in unresectable HCC. Patients received intravenous PD-1 inhibitor 200mg(Camrelizumab, Tislelizumab, or Sintilimab) plus oral Apatinib 250 mg or Lenvatinib 12mg (for bodyweight ≥60 kg) or 8 mg/kg (for bodyweight <60 kg) daily, and additional SFRT for primary liver tumor. PD-1 inhibitor is administered for 2 years or until disease progression or intolerance. Anti-VEGFR is continued until disease progression or intolerance. SFRT implementation plan is as follows: The GTV consists of 2-5 sub-target volumes, which are cylindrical shapes with a diameter of 1.6cm, a height of 2cm, and an interval of 3-5cm. The total volume of the GTV is about 8-20cc, and the distance between the GTV and the OARs is greater than 2cm. The prescribed dosage for each course of radiotherapy is 24 Gy in 3 daily fractions (8Gy x 3F), with a 3-week interval between courses (Q3W). The total courses of radiotherapy shall not be less than 2 (depending on the efficacy and cumulative dose of OARs). The primary endpoint is objective response rate (ORR), and secondary endpoints include overall survival (OS), progression-free survival (PFS), and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. Eastern Cooperative Oncology Group (ECOG) -Performance Status(PS):0-1 points；
3. Patient clinically or pathologically diagnosed with hepatocellular carcinoma；
4. Advanced hepatocellular carcinoma that is inoperable
5. Expected survival period≥3 months;
6. Liver function grade Child-Pugh A or better grade B (7 points);

Exclusion Criteria:

1. Prior invasive malignancy unless disease-free for a minimum of 2 years
2. Prior radiotherapy to the region of the liver that would result in overlap of radiation therapy fields
3. Prior selective internal radiotherapy/ablation, at any time
4. Untreated active hepatitis B or hepatitis C
5. Moderate to severe or intractable ascites
6. Untreated or incompletely treated esophageal or gastric varices
7. Severe, active co-morbidity, defined as follows:

   Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration Myocardial infarction within the last 6 months prior to study entry Acute bacterial or fungal infection requiring intravenous antibiotics within 28 days prior to study entry A bleeding episode within 6 months prior to study entry due to any cause. Thrombolytic therapy within 28 days prior to study entry. Known bleeding or clotting disorder. Uncontrolled psychotic disorder
8. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
9. Prior solid organ transplantation.
10. Immunodeficiency diseases (including HIV) or autoimmune diseases require systemic immunosuppressive therapy (prednisone dosage>10mg per day)
11. Prior or active thrombotic or bleeding disorders, hemoptysis, cerebral vascular accident, significant cardiac disease (ischemic or congestive heart failure), or gastrointestinal perforation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 36 months after registration
  Objective response rate will be ratepresented as a proportion of the total.

SECONDARY OUTCOMES:
Progression-free survival | 36 months after registration
  Progression-free survival and overall survival are evaluated using the Kaplan-Meier curve. Verified through one sample proportion test.
Overall survival | 36 months after registration
  Progression-free survival and overall survival are evaluated using the Kaplan-Meier curve. Verified through one sample proportion test.
Adverse event (Toxicity) | 36 months after registration
  Toxicity will be evaluated using CTCAE version 5.0 and presented as a proportion of the total.
Tumor marker response: AFP | 36 months after registration
  Tumor marker is descriptive as statistics such as mean, standard deviation, and median for continuous data will be presented, and changes in values before and after treatment will be compared and evaluated using paired t-test or Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Yaocan Xu, MD, Principal Investigator — Guiping People's Hospital
Locations (1):
- Guiping People's Hospital, Guiping, Guangxi, China

IPD SHARING:
Plan to Share IPD: No